CLINICAL TRIAL: NCT05901025
Title: Homologous Recombination Repair Pathway Gene Mutation Spectrum in Chinese Breast Cancer Patients: A Multi-center, Prospective, Observational Study
Brief Title: Homologous Recombination Repair Pathway Gene Mutation Spectrum in Chinese Breast Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kunwei Shen, Professor, Director of Comprehensive Breast Health Center, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: RJBC-HRR
Record Dates: First submitted 2023-06-04; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: Homologous Recombination Repair Pathway; Outcome; Mutation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this clinical trial is to learn about the mutation spectrum of homologous recombination repair pathway genes and its instructive significance in the treatment of Chinese breast cancer patients.

DETAILED DESCRIPTION:
The main questions it aims to answer are:

1. What is the mutation spectrum of homologous recombination repair pathway genes in Chinese breast cancer patients?
2. Does homologous recombination repair pathway gene mutation have an impact on patient outcome (breast cancer recurrence, neoadjuvant chemotherapy efficacy, treatment decisions, etc.) ? There is no intervention on participants, but all participants will be given regular follow-up post surgery according to ASCO guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Pathology-confirmed breast cancer patients who meet at least one of the criteria below:

   * Triple-negative breast cancer
   * Age ≤ 50 years
   * Male breast cancer
   * With personal or family history of malignancy: breast cancer, ovarian cancer, prostate cancer, pancreatic cancer, other malignancies
   * HER-2 negative recurrent or metastatic breast cancer
   * HER-2 negative high-risk breast cancer:

   A: Neoadjuvant phase: non-pathological complete response for triple-negative breast cancer; non-pathological complete response AND CPS+EG score ≥ 3 for hormone receptor positive breast cancer B: Adjuvant phase: ≥ pT2 or ≥ pN1 for triple-negative breast cancer; ≥ 4 lymph node metastasis for hormone receptor positive breast cancer
2. Having been or intended to be tested for germline and (or) somatic homologous recombination repair gene mutations
3. Consent to providing medical charts and homologous recombination repair gene testing results, and being cooperative for long-term follow-up

Exclusion Criteria:

1. Homologous recombination repair gene testing results unavailable
2. Other factors deemed by the investigators that may sabotage the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-06-05 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2033-06-30 (Estimated)

PRIMARY OUTCOMES:
Homologous recombination repair pathway gene mutation spectrum | At recruitment
  to reveal the homologous recombination repair pathway gene mutation spectrum

SECONDARY OUTCOMES:
Breast cancer events | At 5 years from surgery
  to compare the incidence of breast cancer-related events and deaths between patients with or without homologous recombination repair pathway gene mutation(s)
Treatment decision and appliance | At 5 years from surgery
  to compare the treatment decision and appliance between patients with or without homologous recombination repair pathway gene mutation(s)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pierce LJ, Levin AM, Rebbeck TR, Ben-David MA, Friedman E, Solin LJ, Harris EE, Gaffney DK, Haffty BG, Dawson LA, Narod SA, Olivotto IA, Eisen A, Whelan TJ, Olopade OI, Isaacs C, Merajver SD, Wong JS, Garber JE, Weber BL. Ten-year multi-institutional results of breast-conserving surgery and radiotherapy in BRCA1/2-associated stage I/II breast cancer. J Clin Oncol. 2006 Jun 1;24(16):2437-43. doi: 10.1200/JCO.2005.02.7888. Epub 2006 Apr 24. PMID 16636335
- [Background] Cao W, Xie Y, He Y, Li J, Wang T, Fan Z, Fan T, Ouyang T. Risk of ipsilateral breast tumor recurrence in primary invasive breast cancer following breast-conserving surgery with BRCA1 and BRCA2 mutation in China. Breast Cancer Res Treat. 2019 Jun;175(3):749-754. doi: 10.1007/s10549-019-05199-8. Epub 2019 Mar 20. PMID 30895535
- [Background] Tutt ANJ, Garber JE, Kaufman B, Viale G, Fumagalli D, Rastogi P, Gelber RD, de Azambuja E, Fielding A, Balmana J, Domchek SM, Gelmon KA, Hollingsworth SJ, Korde LA, Linderholm B, Bandos H, Senkus E, Suga JM, Shao Z, Pippas AW, Nowecki Z, Huzarski T, Ganz PA, Lucas PC, Baker N, Loibl S, McConnell R, Piccart M, Schmutzler R, Steger GG, Costantino JP, Arahmani A, Wolmark N, McFadden E, Karantza V, Lakhani SR, Yothers G, Campbell C, Geyer CE Jr; OlympiA Clinical Trial Steering Committee and Investigators. Adjuvant Olaparib for Patients with BRCA1- or BRCA2-Mutated Breast Cancer. N Engl J Med. 2021 Jun 24;384(25):2394-2405. doi: 10.1056/NEJMoa2105215. Epub 2021 Jun 3. PMID 34081848
- [Background] Tung NM, Robson ME, Ventz S, Santa-Maria CA, Nanda R, Marcom PK, Shah PD, Ballinger TJ, Yang ES, Vinayak S, Melisko M, Brufsky A, DeMeo M, Jenkins C, Domchek S, D'Andrea A, Lin NU, Hughes ME, Carey LA, Wagle N, Wulf GM, Krop IE, Wolff AC, Winer EP, Garber JE. TBCRC 048: Phase II Study of Olaparib for Metastatic Breast Cancer and Mutations in Homologous Recombination-Related Genes. J Clin Oncol. 2020 Dec 20;38(36):4274-4282. doi: 10.1200/JCO.20.02151. Epub 2020 Oct 29. PMID 33119476
- [Background] Telli ML, Jensen KC, Vinayak S, Kurian AW, Lipson JA, Flaherty PJ, Timms K, Abkevich V, Schackmann EA, Wapnir IL, Carlson RW, Chang PJ, Sparano JA, Head B, Goldstein LJ, Haley B, Dakhil SR, Reid JE, Hartman AR, Manola J, Ford JM. Phase II Study of Gemcitabine, Carboplatin, and Iniparib As Neoadjuvant Therapy for Triple-Negative and BRCA1/2 Mutation-Associated Breast Cancer With Assessment of a Tumor-Based Measure of Genomic Instability: PrECOG 0105. J Clin Oncol. 2015 Jun 10;33(17):1895-901. doi: 10.1200/JCO.2014.57.0085. Epub 2015 Apr 6. PMID 25847929
- [Background] Silver DP, Richardson AL, Eklund AC, Wang ZC, Szallasi Z, Li Q, Juul N, Leong CO, Calogrias D, Buraimoh A, Fatima A, Gelman RS, Ryan PD, Tung NM, De Nicolo A, Ganesan S, Miron A, Colin C, Sgroi DC, Ellisen LW, Winer EP, Garber JE. Efficacy of neoadjuvant Cisplatin in triple-negative breast cancer. J Clin Oncol. 2010 Mar 1;28(7):1145-53. doi: 10.1200/JCO.2009.22.4725. Epub 2010 Jan 25. PMID 20100965
- [Background] Isakoff SJ, Mayer EL, He L, Traina TA, Carey LA, Krag KJ, Rugo HS, Liu MC, Stearns V, Come SE, Timms KM, Hartman AR, Borger DR, Finkelstein DM, Garber JE, Ryan PD, Winer EP, Goss PE, Ellisen LW. TBCRC009: A Multicenter Phase II Clinical Trial of Platinum Monotherapy With Biomarker Assessment in Metastatic Triple-Negative Breast Cancer. J Clin Oncol. 2015 Jun 10;33(17):1902-9. doi: 10.1200/JCO.2014.57.6660. Epub 2015 Apr 6. PMID 25847936
- [Background] Tutt A, Tovey H, Cheang MCU, Kernaghan S, Kilburn L, Gazinska P, Owen J, Abraham J, Barrett S, Barrett-Lee P, Brown R, Chan S, Dowsett M, Flanagan JM, Fox L, Grigoriadis A, Gutin A, Harper-Wynne C, Hatton MQ, Hoadley KA, Parikh J, Parker P, Perou CM, Roylance R, Shah V, Shaw A, Smith IE, Timms KM, Wardley AM, Wilson G, Gillett C, Lanchbury JS, Ashworth A, Rahman N, Harries M, Ellis P, Pinder SE, Bliss JM. Carboplatin in BRCA1/2-mutated and triple-negative breast cancer BRCAness subgroups: the TNT Trial. Nat Med. 2018 May;24(5):628-637. doi: 10.1038/s41591-018-0009-7. Epub 2018 Apr 30. PMID 29713086
- [Background] Yu KD, Ye FG, He M, Fan L, Ma D, Mo M, Wu J, Liu GY, Di GH, Zeng XH, He PQ, Wu KJ, Hou YF, Wang J, Wang C, Zhuang ZG, Song CG, Lin XY, Toss A, Ricci F, Shen ZZ, Shao ZM. Effect of Adjuvant Paclitaxel and Carboplatin on Survival in Women With Triple-Negative Breast Cancer: A Phase 3 Randomized Clinical Trial. JAMA Oncol. 2020 Sep 1;6(9):1390-1396. doi: 10.1001/jamaoncol.2020.2965. PMID 32789480